CLINICAL TRIAL: NCT05672641
Title: Is Inertial Training More Effective Than Conventional Strength Training?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University in Zielona Góra (Other)
Collaborators: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Mariusz Naczk, professor, University in Zielona Góra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UZielonaGora
Record Dates: First submitted 2022-12-20; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Traditional Strength Training vs Inertial Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inertial training group (Experimental): 13 young men, physical education students. Inertial training was performed three times a week (Monday, Wednesday, Friday, between 7:00 a.m. and 8:30 a.m.) for 6 weeks using Cyklotren device (Inerion, Poland).
  Interventions: Other: Inertial training
- Body building training group (Experimental): 13 young men, physical education students. Body building training was performed three times a week (Monday, Wednesday, Friday, between 7:00 a.m. and 8:30 a.m.) for 6 weeks using traditional free weights.
  Interventions: Other: Body building training

INTERVENTIONS:
Other: Inertial training — Inertial training group performed their training three times a week (Monday, Wednesday, and Friday) between between 7:00 a.m. and 8:30 a.m. for 6 weeks. Participants performed inertial training using Cyklotren (Inerion, Poland). Before each training session, a standardized warm-up was performed. Each session trained two muscle groups: elbow flexors and knee extensors. Each exercise included 3 sets, with the right and left extremities worked separately. In each set 12 repetitions were performed. A 2-minute break occurred between consecutive sets. Each exercise for elbow flexors was performed in standing position. Each exercise for knee extensors was performed in seated position in a bench. The range of motion for elbow flexors was approximately 130 degrees and for knee extensors was approximately 80 degrees.
  Arms: Inertial training group
Other: Body building training — Body building group performed body building training three times a week (Monday, Wednesday, and Friday) between 7:00 a.m. and 8:30 a.m. for 6 weeks using free weights. Before each training session, a standardized warm-up was performed. Each session trained two muscle groups: elbow flexors and knee extensors. Each exercise included 3 sets, with the right and left extremities worked separately. In each set 12 repetitions were performed. A 2-minute break occurred between consecutive sets. Each exercise for elbow flexors was performed in standing position. Each exercise for knee extensors was performed in seated position in a bench. The range of motion for elbow flexors was approximately 130 degrees and for knee extensors was approximately 80 degrees.
  Arms: Body building training group

SUMMARY:
The data concerning the efficacy of inertial training vs conventional strength training are contradictory. The aim of the study was to compare the impact of inertial training and body building training on elbow flexors and knee extensor strength. Twenty-six young untrained men were randomized to the inertial training (IT; n = 13) or body building group (BBT; n = 13). Both groups performed strength training three times a week for 6; IT - inertial training, BBT - body building training. Each training session included 12 exercise sets involving the elbow flexors and knee and extensors muscles worked separately (3 sets per single muscle group). The training loads were 70% of 1RM for the upper and lower extremities. Before and after training, the maximum force of trained muscles was evaluated under training conditions (one repetition maximum - 1 RM and maximal force under inertial conditions - IFmax) and under isometric conditions (MVT). Moreover, CMJ, SJ, pull-up test, circumferences of the limbs were also evaluated.

DETAILED DESCRIPTION:
A group of 42 young men attended an initial recruitment meeting and all 30 men agreed to participate in the study. The study finally included twenty-six men (mean ± standard deviation: age, 20.4 ± 1.18 years; body mass, 81.0 ± 11.4 kg; height, 184 ± 6.28 cm). The participants were physical education students, but all of them were untrained. The participants were randomly allocated into two groups: inertial training group: IT (n = 13) and a body building training group BBT (n = 13) with the chit method - a simple method of generating random sequence. Both groups participated in 6 weeks of training, IT performed inertial training, BBT performed body building training. All participants were asked to maintain their current level of physical activity and diet throughout the duration of the study. However, we did not control their lifestyle.

Before and after the training muscle strength under different conditions were tested. Moreover, jumping ability, body composition, circumferences of the limbs were evaluated. Each time measurements were performed in five separate days.

1RM

Measurement of 1RM and estimation of training loads. Before training participants were learned techniques of exercise in body building and inertial conditions in two a familiarization sessions. Then, 1RM was determined for the unilateral elbow flexion in standing position using dumbbells and for the unilateral leg extension in sitting position for all participants. 1RM was determined using traditional weights. Next the participants performed 1 set of unilateral flexion in the elbow joint (12 repetitions) and 1 set of unilateral extension in the knee joint with a load of 70% 1RM. During each set, the time of its performance was measured - the participants tried to complete this set in the shortest possible time. Two days later, the training load for inertial training was determined using Cyklotren (Inerion, Poland). Each participant performed several sets of exercises with different loads. The load was increased/decreased so that the performance time of 12 repetitions (as fast as possible) was the same (with an accuracy of 0.5 s) as in the set time with the 70% 1RM using traditional weights. If in three sets between which 5-minute breaks were applied, it was not possible to determine the load in inertial exercises, the test was repeated on the next day. The range of motion and the body position of the participant during load determination were identical to those in the body-building conditions.

Measurement of maximal force under inertial conditions. The maximal force under inertial conditions (IFmax) was measured using Cyklotren inertial device (Inerion, Poland). Participant position during IFmax measurements both for elbow flexors and knee extensors was the same as during 1RM test. Briefly, after a warm-up, each participant performed a 10-s maximal strength test (elbow flexion and knee extension) the right and left arms separately, with a 2-minute break between measurements. Estimated training loads were used during testing. The range of motion for elbow flexors was approximately 130 degrees and for knee extensors approximately 80 degrees. Cyklotren device displayed on the screen and recorded force level for each repetition, the highest value of force (N) was used for future analysis.

Maximal voluntary torque (MVT) measurement Maximal torque derived from isometric muscle actions were determined using a specialized Biodex 4 Pro device (Shirley, New York, USA). Data collection was preceded by a familiarization session. Biomechanical measurements were collected in a seated position. During elbow flexor measurement one hand grasped the device handle as the other remained on the abdomen. The shoulder joint and elbow joint of active arm was set at 90° flexion. During knee extensor measurement the ankle of the active leg was attached to the Biodex moving shin. In the starting position, the thigh of the dominant leg was immobilized at 90° in relation to the trunk, and the knee was also positioned at 90°. In order to eliminate the activity of undesired muscle groups, the participant's trunk was stabilized using belts across the chest. Prior to the measurements, participants were given verbal instructions on the experiment's design. Each of the participants performed three maximal isometric contractions (for each tested muscle group for both upper and lower extremities), each lasting 3 s separated 30 s. breaks. The highest value among the three trials was adopted for further analysis.

Jump tests The vertical jump tests required each participant to perform three SJ with a 30s passive rest period between each effort, followed by three CMJ with a 30s passive rest period between each effort. Both the SJ and CMJ were performed using TENDO JumpMat (Trencin, Slovakia). The highest value of jump (cm) among the three trials was adopted for further analysis.

Upper limbs strength - pull-ups. Participant grasped an overhead horizontal bar with a shoulder width, with a supinated forearm position, while hanging vertically (with feet just above the ground). The body was pulled upright in a linear path until the underside of the chin achieved level with or above the top surface of the horizontal bar. The participants had to avoid all swinging, kicking, and twisting motions. Each participant had to perform as many repetitions as possible.

Body composition To evaluate the influence of training on body composition, bioelectrical impedance device (Tanita MC-980 MA, Tanita Corporation, Tokyo, Japan) was used. The participants were asked to maintain a normal state of hydration prior to measurement, and they were not allowed to exercise, or eat for 12 h preceding the measurements. The measurements were made in the morning, according to manufacturer's guidelines.

Circumferences of the limbs Circumferences of the upper arm were measured at the largest part of the limb in the tensed muscle. The thigh circumference was determined at the half length of the loaded limb. The same person took every measurement to the nearest 0.5 cm three times. The mean value of the three measurements was used to future calculation.

ELIGIBILITY:
Inclusion Criteria:

* lack of regular training prior 24 months well health status, having a current Covid 19 vaccination certificate could participate in the study

Exclusion Criteria:

* tendon or ligament injury in the prior 2 months, fractures in the prior 3 months

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2022-12-18 (Actual)

PRIMARY OUTCOMES:
Elbow flexors and knee extensors strength under traditional free weights conditions. | 6 weeks
  Elbow flexors and knee extensors strength under traditional free weights conditions was tested. Before testing, a standardized warm-up comprising 5 minutes of submaximal cycling on the lower and upper body ergometer and eight repetitions with about 50% 1RM was performed. 1RM was determined for the unilateral elbow flexion in standing position using dumbbells and for the unilateral leg extension in sitting position for all participants. 1RM was determined using traditional weights. Participants increased the load attempting their 1RM. A series of single attempts were completed until a 1RM is achieved. Rest periods were 2 minutes between each single attempt. 1RMs were achieved within 3-7 attempts.
Elbow flexors and knee extensors strength under inertial conditions. | 6 weeks
  The maximal force under inertial conditions (IFmax) was measured using Cyklotren inertial device (Inerion, Poland). IFmax was determined for the unilateral elbow flexion in standing position using Cyklotren and for the unilateral leg extension in sitting position using Cyklotren for all participants. Briefly, after a warm-up, each participant performed a 10-s maximal strength test (elbow flexion and knee extension) the right and left arms separately, with a 2-minute break between measurements. Estimated training loads were used during testing. The range of motion for elbow flexors was approximately 130 degrees and for knee extensors approximately 80 degrees. Cyklotren device displayed on the screen and recorded force level for each repetition, the highest value of force (N) was used for future analysis.
  Description of training loads estimation. Under free weights conditions all the participants performed 1 set of unilateral flexion in the elbow joint (12 repetitions) and 1 set of

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zielona Gora, Zielona Góra, Poland